CLINICAL TRIAL: NCT01049048
Title: The Effect of Vitamin D Statues on Endothelial Function
Acronym: CVD Cookie
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: H-2008-0190
Record Dates: First submitted 2010-01-12; First posted 2010-01-14 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2011-03

CONDITIONS: Cardiovascular Diseases; Vitamin D Deficiency
Keywords: Endothelial Function; Arterial stiffness; Vitamin D
MeSH Terms: conditions — Cardiovascular Diseases; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): This group receives placebo chocolate cookies with no vitamin D3 added.
  Interventions: Dietary Supplement: Placebo
- Vitamin D3 (Experimental): This group receives 2500 IU of Vitamin D3 added to a chocolate cookie daily.
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — 2500 IU Vitamin D3
  Arms: Vitamin D3
Dietary Supplement: Placebo — No (0 IU) vitamin D3 added to cookie.
  Arms: Control

SUMMARY:
In the United States, cardiovascular disease causes over one-third of all deaths and vitamin D deficiency is an epidemic. An increasing body of data suggests that low vitamin D status adversely impacts the cardiovascular system. It is our fundamental hypothesis that vitamin D deficiency is a risk factor for cardiovascular disease by causing endothelial dysfunction. Moreover, we hypothesize that vitamin D supplementation will restore endothelial function, thereby reducing cardiovascular disease risk.

This pilot research will be conducted in 64 post-menopausal women participating in an existing study of vitamin D supplementation (32 will receive vitamin D3 2,500 IU daily, the others matching placebo) and will explore the effects of vitamin D on endothelial function and arterial reactivity. Post-menopausal women aged 55-65 years are chosen due to their highest risk for development of a subsequent new cardiovascular disease diagnosis. All study participants will have fasting laboratory and noninvasive vascular ultrasound studies performed at baseline and four months later. The primary outcome measure of this pilot study is change in markers of endothelial function and arterial stiffness with vitamin D3 therapy. If our hypotheses are correct, our long-term goals include investigation of the effect of vitamin D repletion on subclinical atherosclerosis and subsequent cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, community-dwelling ambulatory post-menopausal women.
* Able and willing to sign informed consent.
* Ages: 55-65.
* Baseline serum 25OHD concentration > 10 ng/ml and < 60 ng/ml
* Not pregnant
* Willing to avoid use of cod-liver oil and non-study vitamin D supplementation; standard multiple vitamins containing ≤ 400 IU used no more than once daily will be allowed.
* Willing to utilize sunscreen of SPF-15 or higher when sun exposure for more than 15 minutes is expected.
* Willing to fast for 12 hours.

Exclusion Criteria:

* Current hypercalcemia (serum calcium > 10.5 mg/dl) or untreated primary hyperparathyroidism.
* History of nephrolithiasis
* Baseline 24-hour urine calcium > 250 mg
* Known risk factors for hypercalcemia, e.g., malignancy, tuberculosis, sarcoidosis, Paget's disease.
* History of any form of cancer within the past five years with the exception of adequately treated squamous cell or basal cell skin carcinoma.
* Known previous personal history of cardiovascular disease.
* Renal failure; defined as a calculated creatinine clearance (using the Cockroft-Gault approach) of ≤ 25 ml/minute.
* Severe end-organ disease, e.g., cardiovascular, hepatic, hematologic, pulmonary, etc., which might limit the ability to complete this study.
* Treatment with any drug known to interfere with vitamin D metabolism, e.g., phenytoin, phenobarbital.
* Known malabsorption syndromes, e.g., celiac disease, active inflammatory bowel disease, etc.
* Known allergy to chocolate.
* Use of medications known to alter bone turnover including bisphosphonates, estrogen, selective estrogen receptor modulators, parathyroid hormone, testosterone or calcitonin.
* Treatment with any active metabolites of vitamin D, e.g., calcitriol, within six months of screening.
* Use of tanning beds or salons or unwillingness to utilize sunscreen during periods of sun exposure of 15 minutes or longer.

Ages: 55 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure of this pilot study is change in markers of endothelial function and arterial stiffness with vitamin D3 therapy. | 17 months

CONTACTS AND LOCATIONS:
Overall Officials: Rekha Ramamurthy, M.D., Principal Investigator — University of Wisconsin Osteoporosis Clinical Center and Research Program; Neil C Binkley, M.D., Study Director — University of Wisconsin Osteoporosis Clinical Center and Research Program
Locations (1):
- University of Wisconsin Osteoporosis Clinical and Research Program, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Gepner AD, Ramamurthy R, Krueger DC, Korcarz CE, Binkley N, Stein JH. A prospective randomized controlled trial of the effects of vitamin D supplementation on cardiovascular disease risk. PLoS One. 2012;7(5):e36617. doi: 10.1371/journal.pone.0036617. Epub 2012 May 7. PMID 22586483